CLINICAL TRIAL: NCT04033354
Title: A Randomized, Double-Blind, Multicenter, Phase III Clinical Study of HLX10 (Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection) + Chemotherapy (Carboplatin Nanoparticle Albumin Bound (Nab)-Paclitaxel) vs Chemotherapy (Carboplatin Nab-Paclitaxel) as First-Line Therapy for Locally Advanced or Metastatic Squamous Non Small Cell Lung Cancer (NSCLC)
Brief Title: A Randomized, Double-blind, Placebo Controlled Phase III Study to Investigate Efficacy and Safety of First-Line Treatment With HLX10 + Chemotherapy (Carboplatin-Nanoparticle Albumin Bound (Nab) Paclitaxel) in Patients With Stage IIIB/IIIC or IV NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-004-NSCLC303
Record Dates: First submitted 2019-07-19; First posted 2019-07-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Squamous Non Small Cell Lung Cancer
Keywords: Locally Advanced or Metastatic; Squamous Non Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Carboplatin; Taxes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): HLX10 + chemotherapy (carboplatin nab paclitaxel)
  Interventions: Drug: HLX10; Drug: carboplatin and nab paclitaxel
- B (Placebo Comparator): Placebo + chemotherapy (carboplatin nab paclitaxel), After 1st PD, the subject will be unblinded by the investigator and be continued with HLX10 monotherapy
  Interventions: Drug: carboplatin and nab paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: HLX10 — HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  Arms: A
Drug: carboplatin and nab paclitaxel — chemotherapeutics
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
This study is a randomized, double-blind, multicenter, phase III clinical study to compare the clinical efficacy and safety of HLX10 + chemotherapy vs chemotherapy in subjects with locally advanced or metastatic squamous NSCLC who have not previously received systemic treatment.

Eligible subjects in this study will be randomized to Arm A or Arm B at 2:1 ratio as follows:

Arm A (HLX10 arm): HLX10 + chemotherapy (carboplatin nab paclitaxel) Arm B (placebo arm): Placebo + chemotherapy (carboplatin nab paclitaxel) The three stratification factors for randomization include: PD-L1 expression level (Tumor Proportion Scores [TPS]≥50%, 50%>TPS≥1%, TPS<1%), Asian population (yes or no), NSCLC stage (stage IIIB/IIIC or stage IV), and carboplatin AUC (5 or 6).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed stage IIIB/IIIC and stage IV (AJCC Edition 8) squamous NSCLC where surgery or radiotherapy cannot be performed.
2. No known sensitizing EGFR mutations or ALK, ROS1 gene rearrangements.
3. Major organs are functioning well
4. Participant must keep contraception
5. Patients with prior denosumab use who can agree to switch to bisphosphonate therapy for bone metastases in the study.

Exclusion Criteria:

1. Patients with histologically non-squamous NSCLC. Mixed tumors will be classified according to the primary cell type. Patients do not meet the requirements for enrollment if small cell components and neuroendocrine carcinoma components are present. For non-small cell histology, patients meet the requirements for enrollment if squamous components (e.g., adenosquamous) are present.
2. Patients with known history of severe hypersensitivity to any monoclonal antibody.
3. Patients with known hypersensitivity to any compositions of carboplatin or nab-paclitaxel.
4. Pregnant or breastfeeding females.
5. Patients with a known history of psychotropic drug abuse or drug addiction; or a history of alcohol abuse.
6. Patients who have other factors that could lead to the early termination of this study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
tumor assessment | Baseline until disease progression or death, whichever occurs first (up to approximately 24months)
  Progression-free survival (PFS) (assessed by the independent radiology review committee [IRRC] based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)

CONTACTS AND LOCATIONS:
Locations (92):
- Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia, United States
- China (53):
  - Anhui Medical University - The Second Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Army Medical University,PLA, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Fuzhou Pulmonary hospital of Fujian, Fuzhou, Fujian
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Fifth Affiliared Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University - Tumor Hospital (The Third Affiliated Hospital), Harbin, Heilongjiang
  - The fourth affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-japan union hospital of jilin university, Changchun, Jilin
  - Jilin Province Cancer Hospital, Changchun, Jilin
  - Jilin Province People's Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - The second Hospital of Jilin University, Changchun, Jilin
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital - Internal Medicine, Jinan, Shandong
  - Linyi City People Hospital, Linyi, Shandong
  - Shandong Linyi Tumor Hospital, Linyi, Shandong
  - Shanghai Eastern Hospital /Affliated Eastern Hospital of Ton, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Yunnan cancer hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
- Georgia (8):
  - High Technology Hospital MedCenter LTD, Batumi
  - JSC Evex Clinics, St.Nikolozi Medical Centre, Kutaisi
  - Acad.F.Todua Medical Center - Research Institute of Clinical Medicine LTD, Tbilisi
  - Institute of Clinical Oncology LTD, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic HELSICORE, Tbilisi
  - Multiprofile Clinic Consilium Medula LTD, Tbilisi
  - New Hospitals LTD, Tbilisi
  - Scientific Research Center of Oncology LTD, Tbilisi
- Poland (2):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Wojew. Wielospecjalistyczne Centrum Onkologii i Traumatologi, Lodz
- Russia (9):
  - LLC "VitaMed ", Moscow
  - University Clinic of Headaches, Moscow
  - Budgetary Healthcare Institution of Omsk Region "C, Omsk
  - GBUZ Orenburg Regional Clinical Oncology Dispensar, Orenburg
  - First St. Petersburg State Medical University n. a. Pavlov, Saint Petersburg
  - Limited Liability Company "AV Medical Group", Saint Petersburg
  - LLC - Strategic Medical systems - Oncology - Oncology, Saint Petersburg
  - PMI "Evromedservice", Saint Petersburg
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- Turkey (Türkiye) (10):
  - Ankara University Medical Faculty - Oncology, Ankara
  - Hacettepe University Medical Faculty - Medical Oncology, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Medipol Mega Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Izmir Medical Park Hospital - Medical Oncology, Izmir
  - Kocaeli University Research and Practice Hospital, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Inonu University Turgut Ozal Medical Center, Malatya
- Ukraine (9):
  - Komunalna ustanova "Chernivets, Chernivtsi
  - Komunalnyi zaklad Miska bahato, Dnipro
  - Komunalne nekomertsiine pidpry, Kharkiv
  - PE PMC "Acinus", Kirovohrad
  - Medychnyi tsentr "Mriya Med-Servis", Kryvyi Rih
  - Limited Liability Company "Medical Center "Verum", Kyiv
  - Komunalne pidpryiemstvo "Volynskyi oblasnyi medychnyi tsentr onkolohii" Volynskoyi oblasnoyi rady, Lutsk
  - Medychnyi tsentr "Onkolaif" LL, Zaporizhzhia
  - Zaporozhye Regional Clinical O, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou C, Hu Y, Arkania E, Kilickap S, Ying K, Xu F, Wu L, Wang X, Viguro M, Makharadze T, Sun H, Luo F, Shi J, Zang A, Pan Y, Chen Z, Jia Z, Kuchava V, Lu P, Zhang L, Cheng Y, Kang W, Wang Q, Yu H, Li J, Zhu J; ASTRUM-004 Investigators. A global phase 3 study of serplulimab plus chemotherapy as first-line treatment for advanced squamous non-small-cell lung cancer (ASTRUM-004). Cancer Cell. 2024 Feb 12;42(2):198-208.e3. doi: 10.1016/j.ccell.2023.12.004. Epub 2024 Jan 4. PMID 38181795